CLINICAL TRIAL: NCT06560788
Title: Chiari II Brain Malformation: The Role of Cerebrospinal Fluid in Neurodevelopmental Defects Associated With Spina Bifida
Brief Title: The Role of CSF in Chiari II Brain Malformation
Status: Not yet recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other); University College London Hospitals (Other)
Responsible Party: Principal Investigator, Amparo Saenz, PhD student and pediatric neurosurgeon, University College, London
Other Study IDs: 23DD12; 344434 (Other: IRAS Number); Z6364106/2024/08/97 (Other: UCL Data Protection registration number)
Record Dates: First submitted 2024-08-12; First posted 2024-08-19 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Myelomeningocele; Brain Malformation; Chiari Malformation Type 2
Keywords: myelomeningocele; Chiari type 2; brain malformations; cognitive impairment; cerebrospinal fluid
MeSH Terms: conditions — Meningomyelocele; Arnold-Chiari Malformation; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Case group 1: Children with Open Spina Bifida and Chiari II Malformation: CSF will be collected during postnatal surgical repair at Great Ormond Street Hospital (GOSH)
  Interventions: Other: collection of cerebrospinal fluid
- Control group 1: Newborns with hydrocephalus undergoing shunt surgery, unrelated to spina bifida: CSF will be collected during suregry at GOSH
  Interventions: Other: collection of cerebrospinal fluid
- Control group 1bis: Infants undergoing spinal surgery for conditions other than SB: CSF will be collected during surgery at GOSH.
  Interventions: Other: collection of cerebrospinal fluid
- Case group 2: Fetuses Undergoing Prenatal Surgery for Spina Bifida: CSF will be collected during prenatal surgery at University College London Hospitals (UCLH).
  Interventions: Other: collection of cerebrospinal fluid
- Control group 2: Aborted fetuses within the gestational age range of 22-24 weeks,: CSF will be collected from fetuses provided by the Human Developmental Biology Resource (HDBR).
  Interventions: Other: collection of cerebrospinal fluid
- Case group 3: mouse model of spina bifida (Cdx2Cre x Pax3flox): CSF will be collected
  Interventions: Other: collection of cerebrospinal fluid
- Control group 3: normal (wild-type) mice: CSF will be collected
  Interventions: Other: collection of cerebrospinal fluid

INTERVENTIONS:
Other: collection of cerebrospinal fluid — CSF is collected as part of routine care in any of the surgeries listed in the control or cases groups. We will take part of that CSF for proteomic analysis

SUMMARY:
Spina bifida, particularly its most severe form known as open spina bifida (myelomeningocele), is a significant congenital disorder that results in profound neurological impairments, including Chiari II malformation. This malformation is associated with the downward displacement of the cerebellum and brainstem into the spinal canal, often leading to hydrocephalus, a condition where cerebrospinal fluid (CSF) accumulates in the brain1. These conditions can result in a range of complications, including cognitive and motor disabilities, learning difficulties, and, in severe cases, early mortality1,2.

While surgical interventions, including prenatal and postnatal surgeries, have been developed to manage the physical manifestations of spina bifida and Chiari II malformation, these procedures have not been fully successful in addressing the associated brain anomalies3. This study aims to explore the hypothesis that the composition of CSF plays a critical role in the development of these brain defects. Specifically, it is hypothesized that the rapid replenishment of CSF, due to its leakage from the open spine in spina bifida, results in a "less mature" fluid composition, which negatively affects neurogenesis and neuronal migration during critical periods of brain development.

DETAILED DESCRIPTION:
Study Population and Methodology

This prospective case-control study will involve the collection of CSF samples from several groups, including:

1. Newborns with open spina bifida undergoing postnatal surgery.
2. Fetuses undergoing prenatal surgery for spina bifida.
3. Newborns with hydrocephalus undergoing shunt surgery (control group).
4. Infants undergoing spinal surgery for conditions unrelated to spina bifida (control group).
5. Age-matched fetuses obtained from the Human Developmental Biology Resource (HDBR) as controls.
6. Mouse models: This includes a genetic mouse model of spina bifida (Cdx2Cre x Pax3flox) and normal (wild-type) mice as controls

These samples will be analyzed using mass spectrometry-based proteomics to identify differences in protein composition and concentrations between the groups. Additionally, brain slices from human embryos and mouse models will be cultured in the presence of these CSF samples to assess the impact on neurogenesis and neuronal migration.

Expected Benefits The findings from this study are expected to provide new insights into the pathogenesis of Chiari II malformation and other associated brain anomalies in children with spina bifida. By understanding how CSF composition influences brain development, the study could pave the way for novel therapeutic strategies aimed at modifying CSF composition during early pregnancy. This could potentially prevent or mitigate the neurological impairments associated with spina bifida, ultimately improving the quality of life for affected individuals.

Impact on Clinical Practice and Policy Should the study confirm the hypothesis, it could lead to changes in clinical practices concerning the management of spina bifida and Chiari II malformation. For instance, it might inform the development of new prenatal treatments or interventions designed to normalize CSF composition before significant brain damage occurs4-6. This would represent a significant advancement in fetal surgery and pediatric neurosurgery, with the potential to influence guidelines and policies within the NHS and other healthcare systems globally.

Relation to Academic Qualification This study is being conducted as part of the Lewis Spitz PhD program at University College London (UCL) and Great Ormond Street Institute of Child Health (GOSH ICH). The research builds upon previous studies sponsored by UCL-ICH/GOSH, particularly those investigating the neurodevelopmental consequences of spina bifida and related congenital conditions.

ELIGIBILITY:
Inclusion Criteria:

Newborns with Spina Bifida (Postnatal Closure)

* Diagnosed with open spina bifida (myelomeningocele).
* Scheduled for postnatal surgical closure of the spinal lesion at Great Ormond Street Hospital (GOSH).
* Age: Between 1 day to 1 year old.

Control Group 1 (Newborns with Hydrocephalus)

* Newborns scheduled for shunt surgery for hydrocephalus unrelated to spina bifida.
* Age and sex matched to the spina bifida newborns as closely as possible.
* Age: Between 1 day to 1 year old.

Control Group 2 (Infants with Spinal Conditions Unrelated to Spina Bifida)

* Infants undergoing paned spinal surgery for conditions such as spinal lipoma, fatty filum, tethered cord, etc.
* Age and sex matched to the spina bifida newborns as closely as possible.
* Age: Between 1 day to 1 year old. Fetuses with Spina Bifida (Prenatal Closure)
* Prenatal diagnosis of spina bifida (myelomeningocele) and scheduled for fetal surgery at UCLH.
* Reviewed by Mr Thompson at his outpatient clinic at GOSH
* Gestational age: Between 22 and 24 weeks.

Control Fetal Samples

* Aborted fetuses within the gestational age range of 22-24 weeks.
* Samples obtained through the Human Developmental Biology Resource (HDBR).

Mouse Models

* Genetic mouse model of spina bifida (Cdx2Cre x Pax3flox).
* At embryonic day (E)13.5 (end of the embryonic period) and E18.5 (just before birth)

Control Mouse Models

* Normal (wild-type) mice to serve as controls.
* Normal brain development
* At embryonic day (E)13.5 (end of the embryonic period) and E18.5 (just before birth)

Exclusion Criteria:

Newborns with Spina Bifida (Postnatal Closure)

* Newborns who have undergone previous surgical intervention.
* Presence of additional unrelated congenital anomalies that could affect cerebrospinal fluid (CSF) composition like meningitis or intraventricular bleeding
* Older than 1 year and 1 month of age.
* Parents refused to participate
* Native language different to English with no translation services available

Control Group 1 (Newborns with Hydrocephalus)

* Newborns with hydrocephalus caused by spina bifida.
* Presence of intraventricular infection or haemorrhage.
* Older than 1 year and 1 month of age.
* Parents refused to participate
* Native language different to English with no translation services available

Control Group 2 (Infants with Spinal Conditions Unrelated to Spina Bifida)

* Infants who were born with spina bifida
* Infants with coexisting conditions that could affect CSF composition like intraspinal tumours, empyema or haemorrhage.
* Older than 1 year and 1 month of age.
* Parents refused to participate
* Native language different to English with no translation services available

Fetuses with Spina Bifida (Prenatal Closure)

* Fetuses with additional major anomalies unrelated to spina bifida like diaphragmatic hernia.
* Gestational age outside the range of 22-24 weeks.
* Surgery performed by other neurosurgery team (not GOSH)
* Parents refused to participate
* Native language different to English with no translation services available

Control Fetal Samples

* Poorly preserved aborted fetuses not suitable for CSF collection.
* Gestational age outside the range 22-24 weeks.

Mouse Models

* Mice with any genetic modifications other than those specified for the spina bifida model.
* Mice with other congenital or acquired anomalies affecting the central nervous system.

Control Mouse Models

● Mice with any genetic modifications or health conditions that could influence the study's outcomes.

Max Age: 1 Year | Sex: All
Age Groups: Child
Study Population: 1. Newborns with open spina bifida undergoing postnatal surgery.
  2. Fetuses undergoing prenatal surgery for spina bifida.
  3. Newborns with hydrocephalus undergoing shunt surgery (control group).
  4. Infants undergoing spinal surgery for conditions unrelated to spina bifida (control group).
  5. Age-matched fetuses obtained from the Human Developmental Biology Resource (HDBR) as controls.
  6. Mouse models: This includes a genetic mouse model of spina bifida (Cdx2Cre x Pax3flox) and normal (wild-type) mice as controls
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Identification of Proteins in Cerebrospinal Fluid (CSF) | 1 year
  The presence of specific proteins in cerebrospinal fluid (CSF) will be identified through proteomic analysis. This outcome will focus on categorizing which proteins are present in the CSF samples from patients with spina bifida and control participants.
Quantification of Protein Concentrations in Cerebrospinal Fluid (CSF) | 1 year
  The concentration of each identified protein in cerebrospinal fluid (CSF) will be measured using proteomic analysis. This outcome will report the amount of each protein present in the CSF, expressed in micrograms per milliliter (µg/mL) or nanograms per milliliter (ng/mL), allowing for comparison between patients with spina bifida and controls.

SECONDARY OUTCOMES:
Measurement of Neurogenesis in Median Ganglionic Eminence (MGE) Cultures | 1 year
  The rate of neurogenesis in the median ganglionic eminence (MGE) of embryonic brain slice cultures will be measured following exposure to cerebrospinal fluid (CSF) from patients with Chiari II malformation and control subjects. The outcome will focus on the number of proliferating neurons per unit area, measured in cells per square millimeter (cells/mm²).
Measurement of Neuronal Migration in Median Ganglionic Eminence (MGE) Cultures | 1 year
  The distance of neuronal migration in the median ganglionic eminence (MGE) of embryonic brain slice cultures will be measured following exposure to cerebrospinal fluid (CSF) from patients with Chiari II malformation and control subjects. The outcome will report the migration distance of neurons, measured in micrometers (µm).

IPD SHARING:
Plan to Share IPD: No
Becuase the infromation provided comes from susceptible (children) population, information won't be shared

REFERENCES:
- [Result] Masse O, Kraft E, Ahmad E, Rollins CK, Velasco-Annis C, Yang E, Warfield SK, Shamshirsaz AA, Gholipour A, Feldman HA, Estroff J, Grant PE, Vasung L. Abnormal prenatal brain development in Chiari II malformation. Front Neuroanat. 2023 Apr 17;17:1116948. doi: 10.3389/fnana.2023.1116948. eCollection 2023. PMID 37139180
- [Result] Schneider J, Mohr N, Aliatakis N, Seidel U, John R, Promnitz G, Spors B, Kaindl AM. Brain malformations and cognitive performance in spina bifida. Dev Med Child Neurol. 2021 Mar;63(3):295-302. doi: 10.1111/dmcn.14717. Epub 2020 Nov 2. PMID 33140418
- [Result] Paslaru FG, Panaitescu AM, Iancu G, Veduta A, Gica N, Paslaru AC, Gheorghiu A, Peltecu G, Gorgan RM. Myelomeningocele Surgery over the 10 Years Following the MOMS Trial: A Systematic Review of Outcomes in Prenatal versus Postnatal Surgical Repair. Medicina (Kaunas). 2021 Jul 12;57(7):707. doi: 10.3390/medicina57070707. PMID 34356988
- [Result] Treble-Barna A, Juranek J, Stuebing KK, Cirino PT, Dennis M, Fletcher JM. Prospective and episodic memory in relation to hippocampal volume in adults with spina bifida myelomeningocele. Neuropsychology. 2015 Jan;29(1):92-101. doi: 10.1037/neu0000111. Epub 2014 Jul 28. PMID 25068670
- [Result] Treble A, Juranek J, Stuebing KK, Dennis M, Fletcher JM. Functional significance of atypical cortical organization in spina bifida myelomeningocele: relations of cortical thickness and gyrification with IQ and fine motor dexterity. Cereb Cortex. 2013 Oct;23(10):2357-69. doi: 10.1093/cercor/bhs226. Epub 2012 Aug 8. PMID 22875857
- [Result] Taylor HB, Barnes MA, Landry SH, Swank P, Fletcher JM, Huang F. Motor contingency learning and infants with Spina Bifida. J Int Neuropsychol Soc. 2013 Feb;19(2):206-15. doi: 10.1017/S1355617712001233. Epub 2013 Jan 8. PMID 23298791
- [Result] David AL. Improving motor function in fetal surgery for open spina bifida. BJOG. 2024 May;131(6):768. doi: 10.1111/1471-0528.17730. Epub 2023 Nov 30. No abstract available. PMID 38037518
- [Result] Vergote S, Van der Stock J, Kunpalin Y, Bredaki E, Maes H, Banh S, De Catte L, Devlieger R, Lewi L, Devroe S, Spencer R, David A, De Vloo P, Van Calenbergh F, Deprest JA. Patient empowerment improves follow-up data collection after fetal surgery for spina bifida: institutional audit. Ultrasound Obstet Gynecol. 2023 Oct;62(4):565-572. doi: 10.1002/uog.26230. Epub 2023 Aug 27. PMID 37099513
- [Result] Bueno D, Parvas M, Nabiuni M, Miyan J. Embryonic cerebrospinal fluid formation and regulation. Semin Cell Dev Biol. 2020 Jun;102:3-12. doi: 10.1016/j.semcdb.2019.09.006. Epub 2019 Oct 12. PMID 31615690
- [Result] Zappaterra MD, Lisgo SN, Lindsay S, Gygi SP, Walsh CA, Ballif BA. A comparative proteomic analysis of human and rat embryonic cerebrospinal fluid. J Proteome Res. 2007 Sep;6(9):3537-48. doi: 10.1021/pr070247w. Epub 2007 Aug 16. PMID 17696520
- [Result] Pal K, Sharma U, Gupta DK, Pratap A, Jagannathan NR. Metabolite profile of cerebrospinal fluid in patients with spina bifida: a proton magnetic resonance spectroscopy study. Spine (Phila Pa 1976). 2005 Feb 1;30(3):E68-72. doi: 10.1097/01.brs.0000152161.08313.04. PMID 15681999
- [Result] Shokohi R, Nabiuni M, Irian S, Miyan JA. In Vitro Effects of Wistar Rat Prenatal and Postnatal Cerebrospinal Fluid on Neural Differentiation and P roliferation of Mesenchymal Stromal Cells Derived from Bone Marrow. Cell J. 2018 Jan;19(4):537-544. doi: 10.22074/cellj.2018.4130. Epub 2017 Nov 4. PMID 29105387
- [Result] Alonso MI, Lamus F, Carnicero E, Moro JA, de la Mano A, Fernandez JMF, Desmond ME, Gato A. Embryonic Cerebrospinal Fluid Increases Neurogenic Activity in the Brain Ventricular-Subventricular Zone of Adult Mice. Front Neuroanat. 2017 Dec 19;11:124. doi: 10.3389/fnana.2017.00124. eCollection 2017. PMID 29311854
- [Result] Eid L, Lachance M, Hickson G, Rossignol E. Ex Utero Electroporation and Organotypic Slice Cultures of Embryonic Mouse Brains for Live-Imaging of Migrating GABAergic Interneurons. J Vis Exp. 2018 Apr 20;(134):57526. doi: 10.3791/57526. PMID 29733310